CLINICAL TRIAL: NCT01591538
Title: Prevalence Study Evaluating the Acquisition of Carriage of Resistant Bacteria in the Gut Flora in Volunteers From French Armed Forces Coming Back From External Operations
Brief Title: Multi-Antibiotic Resistance Carriage in Gut Flora
Acronym: MARC
Status: Completed | Type: Observational
Sponsor: Da Volterra (Industry)
Responsible Party: Sponsor
Other Study IDs: DAV148-EPI-01; ID RCB number : 2011-A01569-32 (Other: AFSSAPS)
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Intestinal Bacteria Flora Disturbance
Keywords: Prevalence; MDRGNB; Acquisition; Middle stay; Endemic area

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lifestyle condition

SUMMARY:
Prevalence Study evaluating the acquisition of carriage of multidrug-resistant Gram-negative bacteria (MDRGNB) in the gut flora in volunteers of French Armed Forces staying from 4 to 6 months outside France.

DETAILED DESCRIPTION:
Emergence of MDRGN bacteria is blowing worldwide up leading to therapeutical failure in hospitalized patients with severe infections, as well as in outpatients with community-acquired infections such as UTI. Variation in prevalence exists across countries and regions. Travels outside own country of residence, like France, whatever the duration (short or long)or the reason (professional or leisure), are known risk factors for acquiring and disseminating MDRGN bacteria. Digestive carriage of multidrug-resistant Enterobacteriaceae could be a source of infection for the host as well as a source of dissemination. Qualitative and quantitative gut colonization by MDRGNB is poorly studied in non-hospitalized people who stayed for a few months out of France. The total amount of multidrug-resistant Enterobacteriaceae influences the spread of the dissemination. In our knowledge, no clinical study has been carried out to qualify and quantify gut colonization by MDRGNB in volunteers after staying 4-6 months outside country of residence such as France. A specific microbiological method will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18 years
* Have given an informed consent by signing the written consent
* Being able to give a stool sample
* Being member of military forces, supported medically by the French Military Health Services (SSA), and to participate outside mission during 4- 6 months

Exclusion Criteria:

* Participating in another biomedical study during the study
* Volunteer unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers from French Armed Forces
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Frequency of MDRGNB (ESBLs or carbapenemases) colonization in gut flora of volunteers after staying 4-6 months outside France | 12 months

SECONDARY OUTCOMES:
Quantitative measurement of MDRGNB in fecal samples (expressed as log10 and percentage) of volunteers after staying 4-6 months outside France | 12 months
Quantitative variation of MDRGNB between the departure and return in volunteers | 12 months
PCR and sequencing of resistance genes from strains of interest | 12 months
Evaluation of risk factors for acquiring MDRGNB in gut flora of volunteers after staying 4-6 months outside France | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste MEYNARD, MD/PhD, Principal Investigator — French Armed Forces
Locations (1):
- Centre d'épidémiologie et de santé publique des armées, Saint-Mandé, France